CLINICAL TRIAL: NCT06957847
Title: Clinical Validation Of The Brachial Blood Pressure Measuring Device Withings BPM Pro 2 According To "The Universal Protocol For The Validation Of Blood Pressure Measuring Devices By The Association For The Advancement Of Medical Instrumentation / European Society Of Hypertension / International Organization For Standardization (AAMI/ESH/ISO) (And Its Amendment 1 (2020) And 2 (2024))" In The General Population.
Brief Title: Clinical Validation of the Blood Pressure Measuring Device Withings BPM Pro 2 (WIHYP-GP)
Acronym: WIHYP-GP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Withings (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2025-A00050-49
Record Dates: First submitted 2025-05-02; First posted 2025-05-05 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Blood Pressure Determination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All patients (Experimental): Patients consenting to participate to the study and compliant to the inclusion criteria
  Interventions: Device: Blood pressure measurement

INTERVENTIONS:
Device: Blood pressure measurement — The patient will be measured alternatively with a reference mercury sphygmomanometer (four times) and the device under study (3 times)

SUMMARY:
The aim of the study is to assess the accuracy of the automatic oscillometric BP measuring device at the brachial level, the WITHINGS BPM Pro 2, in the general population

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years;
* Patient who signed the informed consent form;
* Patient followed-up at site (in-patient or out-patient);
* Patient with arm circumference between 22 cm and 42 cm.

Exclusion Criteria:

* Patient unable to give a consent or understand properly protocol information;
* Patient suffering from arrhythmia;
* Patient with poor quality of Korotkov sounds;
* Patient for whom K5 sounds are absent;
* Patient wearing an implantable electric medical device (pacemaker,…);
* Patient with both upper arms suffering from open wound and/or damaged skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Blood pressure measurement performance evaluation per measure | The time frame is three months.
  The blood pressure (systolic and diastolic blood pressure) measurement performance will be established using the mean value of the differences and the standard deviation between the device under study and the reference for each measure.
Blood pressure measurement performance evaluation by subject | The time frame is three months.
  The blood pressure measurement performance by subject will be established using the mean value of the differences and the standard deviation between the averaged per subject value of blood pressure (systolic and diastolic blood pressure) device under study and its reference.

SECONDARY OUTCOMES:
Safety use of the device | The time frame is three months.
  The rate of adverse effects.

CONTACTS AND LOCATIONS:
Locations (1):
- N2, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: No